CLINICAL TRIAL: NCT04078152
Title: An Open-Label, Multi-Center, Global Study to Evaluate Long Term Safety and Efficacy in Patients Who Are Receiving or Who Previously Received Durvalumab in Other Protocols (WAVE)
Brief Title: Durvalumab Long-Term Safety and Efficacy Study
Acronym: WAVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry); Parexel (Industry); Medidata Solutions (Industry); CISCRP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D910FC00001; 2019-001402-20 (EudraCT Number)
Record Dates: First submitted 2019-08-09; First posted 2019-09-04 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumor
Keywords: non-small cell lung cancer (NSCLC); urothelial cancer; durvalumab; long-term safety, efficacy; overall survival; immunotherapy; checkpoint inhibitor; PD-L1; retreatment; Gastric adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Masking Description: All involved know the identity of the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Durvalumab Monotherapy
  Interventions: Drug: Durvalumab
- Off Treatment (No Intervention): Follow up Only

INTERVENTIONS:
Drug: Durvalumab — IV infusion q4w with 1500mg durvalumab until progressive disease
  Other Names: MEDI4736
  Arms: Treatment

SUMMARY:
The aims of the study are to monitor the long-term safety of durvalumab, to provide continued treatment or retreatment with durvalumab to eligible patients, and to collect overall survival (OS) information.

DETAILED DESCRIPTION:
This is a multicenter, open-label, global study that will enroll patients who are currently receiving durvalumab monotherapy, or have previously received durvalumab as monotherapy or in combination with any other approved or investigational anticancer agents, in an eligible AstraZeneca/MedImmune-sponsored clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 18 years or older, at the time of signing the ICF. For subjects aged < 20 years and enrolled in Japan, a written ICF should be obtained from the subject and his or her legally acceptable representative.
2. Patient received durvalumab monotherapy and/or durvalumab containing combination in an AstraZeneca/MedImmune-sponsored parent clinical study that is approved for enrollment into this study.
3. Patients who received durvalumab in combination with any other approved or investigational anticancer agents in the parent clinical study must have completed or discontinued all other anticancer therapy (beyond durvalumab regimen).
4. Patient must be willing and able to provide written informed consent and to comply with scheduled visits and other study procedures.

Exclusion Criteria:

The following exclusion criteria apply only to patients receiving treatment or retreatment:

1. Currently receiving treatment in another interventional study other than the parent clinical study or, for retreatment patients, received treatment during the follow up period with an agent other than durvalumab
2. Any concurrent chemotherapy, IP, biologic or hormonal therapy for cancer treatment
3. Experienced an immune-mediated or non-immune-mediated toxicity that led to permanent discontinuation of durvalumab in parent clinical study
4. Diagnosis of a new primary malignancy since enrollment into the parent clinical study

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (104):
- United States (12):
  - Research Site, Fullerton, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Augusta, Georgia
  - Research Site, Baltimore, Maryland
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Mineola, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Huntersville, North Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
- Research Site, Rosario, Argentina
- Australia (2):
  - Research Site, Box Hill
  - Research Site, Melbourne
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Kortrijk
  - Research Site, Leuven
- Brazil (4):
  - Research Site, Florianópolis
  - Research Site, Ijuí
  - Research Site, Porto Alegre
  - Research Site, São José do Rio Preto
- Research Site, Sofia, Bulgaria
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Toronto, CA
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Newmarket, Ontario
- Research Site, Santiago, Chile
- Research Site, Olomouc, Czechia
- France (3):
  - Research Site, Brest
  - Research Site, Lille
  - Research Site, Lyon
- Germany (2):
  - Research Site, Dresden
  - Research Site, Hanover
- Research Site, Holargos, Athens, Greece
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Miskolc
- Research Site, Chennai, India
- Research Site, Haifa, Israel
- Japan (16):
  - Research Site, Bunkyō City
  - Research Site, Fukushima
  - Research Site, Isehara-shi
  - Research Site, Izumi-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kōtoku
  - Research Site, Nagaoka-shi
  - Research Site, Nagoya
  - Research Site, Natori-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Saga
  - Research Site, Suita-shi
  - Research Site, Sunto-gun
  - Research Site, Tokushima
  - Research Site, Yokohama
- Research Site, Kuching, Malaysia
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Arnhem
- Poland (2):
  - Research Site, Lodz
  - Research Site, Olsztyn
- Romania (2):
  - Research Site, Craiova
  - Research Site, Suceava
- Russia (5):
  - Research Site, Arkhangelsk
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, pos.Pesochnyi
  - Research Site, Saint Petersburg
- Research Site, Kamenitz, Serbia
- South Korea (6):
  - Research Site, Daegu
  - Research Site, Gwangju
  - Research Site, Gyeongsangnam-do
  - Research Site, Seogu
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (8):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Jaén
  - Research Site, Madrid
  - Research Site, Marbella
  - Research Site, Málaga
  - Research Site, Valencia
- Switzerland (2):
  - Research Site, Bellinzona
  - Research Site, Lausanne
- Taiwan (4):
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Songkhla
- Turkey (Türkiye) (2):
  - Research Site, Adana
  - Research Site, Istanbul
- Ukraine (9):
  - Research Site, Chernivtsі
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kirovohrad
  - Research Site, Kryvyi Rih
  - Research Site, Kyiv
  - Research Site, Sumy
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
- United Kingdom (2):
  - Research Site, London
  - Research Site, Manchester
- Research Site, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D910FC00001&attachmentIdentifier=b7d44aa5-4d78-4092-8fc0-b76fe76a81c0&fileName=D910FC00001-CSP_v4_Redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D910FC00001&attachmentIdentifier=0c28a623-3d31-469f-9b63-0200f0df8a66&fileName=D910FC00001-SAP_v2_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D910FC00001&attachmentIdentifier=89671fcd-e198-4fb4-9f13-613cd6907b63&fileName=D910FC00001-CSR_synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase IV, open-label study was conducted at 112 investigational sites across 31 countries in participants who were receiving durvalumab monotherapy and/or those who previously received durvalumab as a monotherapy or in combination with any other approved or investigational anticancer agent in previously enrolled parent study between 05 Sep 2019 and 31 Oct 2022.
Pre-assignment Details: A total of 163 participants were enrolled in this study.
Groups:
- Cohort 1: Durvalumab Continuation: Cohort 1 included participants who had received durvalumab monotherapy or durvalumab combination therapy under the parent clinical study (including those who underwent retreatment per the parent study) who had not clinically progressed and who were eligible to continue durvalumab treatment after completing dosing of all other anticancer agents, including other investigational agents. Participants received durvalumab monotherapy 1500 milligrams (mg) via intravenous (IV) infusion every 4 weeks on Day 1 of each cycle until confirmed progressive disease (PD), unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- Cohort 2: Durvalumab Restart: Cohort 2 included participants who had completed durvalumab monotherapy or combination therapy with any other approved or investigational anticancer agents in a parent study, without confirmed PD during the period of treatment, and who were potentially eligible for retreatment with durvalumab. Participants received durvalumab monotherapy 1500 mg via IV infusion every 4 weeks on Day 1 of each cycle until confirmed PD, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- Cohort 3: No Restart of Durvalumab: Cohort 3 included participants previously treated with durvalumab monotherapy or in combination with any other approved or investigational anticancer agents who were no longer receiving durvalumab and were not eligible to receive retreatment. Participants did not receive any study drug.
Period: Overall Study
Arm/Group | Cohort 1: Durvalumab Continuation | Cohort 2: Durvalumab Restart | Cohort 3: No Restart of Durvalumab
Started | 100 | 25 | 38
Received Treatment in This Study/Within 90 Days Prior Enrolment in This Study(Safety Analysis Set) | 100 | 7 | 2
Completed | 0 | 0 | 0
Not Completed | 100 | 25 | 38
Not completed — Other | 83 | 22 | 25
Not completed — Development of study specific withdrawal criteria | 1 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 1
Not completed — Death | 10 | 2 | 12
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full analysis set included all participants enrolled in the study, regardless of the treatment received.
Groups:
- Cohort 1: Durvalumab Continuation: Cohort 1 included participants who had received durvalumab monotherapy or durvalumab combination therapy under the parent clinical study (including those who underwent retreatment per the parent study) who had not clinically progressed and who were eligible to continue durvalumab treatment after completing dosing of all other anticancer agents, including other investigational agents. Participants received durvalumab monotherapy 1500 mg via IV infusion every 4 weeks on Day 1 of each cycle until confirmed PD, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Durvalumab Continuation | Cohort 2: Durvalumab Restart | Cohort 3: No Restart of Durvalumab | Total
Number analyzed (Participants) | 100 | 25 | 38 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (10.31) | 66.4 (9.30) | 66.1 (9.95) | 65.7 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 7 | 16 | 41
  Male | 82 | 18 | 22 | 122
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 75 | 16 | 21 | 112
  Black or African American | 0 | 1 | 1 | 2
  Asian | 25 | 8 | 16 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 0 | 0 | 9
  Not Hispanic or Latino | 91 | 23 | 37 | 151
  Missing | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was the development of any untoward medical occurrence (other than progression of the malignancy under evaluation) in a participant or clinical study participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. A SAE was an AE occurring during any study phase that fulfilled one or more of the following: resulted in death; was immediately life-threatening; required in-patient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability or incapacity; was a congenital abnormality or birth defect; was an important medical event that jeopardized the participant or required medical treatment to prevent one of the outcomes listed above.
Time Frame: From the time of signing the informed consent form until the follow-up period is completed (90 days after the last dose of durvalumab); approximately 37 months
Population: The Safety analysis set included those participants who received at least 1 dose of durvalumab in this study or enrolled in this study within 90 days of the last dose of durvalumab or durvalumab combination in the respective parent clinical study. The data is from this study only, parent study data is not included in this table.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Durvalumab Continuation | Cohort 2: Durvalumab Restart | Cohort 3: No Restart of Durvalumab
Number analyzed (Participants) | 100 | 7 | 2
Participants
  Any AEs | 85 | 1 | 0
  Any SAEs | 23 | 0 | 0

2. Secondary Outcome: Cohort 2: Overall Response Rate (ORR)
Description: The ORR was defined as the percentage of participants with a confirmed investigator-assessed response of either complete response (CR) or partial response (PR) from the date of re-initiation of treatment with durvalumab monotherapy. Tumor assessments were performed according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1). CR was defined as the disappearance of all target lesions (TLs) since baseline and reduction in short axis diameter to <10 millimeters (mm) for any pathological lymph nodes selected as TLs. PR was defined as at least a 30% decrease in the sum of the diameters of TL, taking as reference the baseline sum of diameter.
Time Frame: Tumor assessments as determined by the Investigator (at least every 12 weeks) until withdrawal of consent, progression or death; approximately 30 months
Population: The Response evaluable analysis set included those participants who underwent retreatment with durvalumab in Cohort 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Durvalumab Restart
Number analyzed (Participants) | 2
percentage of participants | 0 [0 to 84]

3. Secondary Outcome: Cohort 2: Duration of Response (DOR)
Description: The DOR was defined as the time from first documented CR or PR to time of first documented disease progression or death in the absence of disease progression. Tumor assessments were performed according to RECIST v1.1.
Time Frame: as for outcome 2
Population: The Response evaluable analysis set included those participants who underwent retreatment with durvalumab in Cohort 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2: Durvalumab Restart
Number analyzed (Participants) | 2
months | NA [NA to NA] — As no participant in the response evaluable analysis set was assessed to have had either CR or PR, the DOR analysis was not applicable.

4. Secondary Outcome: Number of Participants Who Were Alive
Description: Number of participants who were alive are reported in this outcome measure. Any participant not known to have died at the time of analysis was censored based on the last recorded date on which the participant was known to be alive.
Time Frame: Up to approximately 37 months
Population: The Full analysis set included all participants enrolled in the study, regardless of the treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Durvalumab Continuation | Cohort 2: Durvalumab Restart | Cohort 3: No Restart of Durvalumab
Number analyzed (Participants) | 100 | 25 | 38
Participants | 90 | 23 | 26

ADVERSE EVENTS:
Time Frame: From the time of signing the informed consent form until the follow-up period is completed (90 days after the last dose of durvalumab); approximately 37 months
Description: The Safety analysis set included those participants who received at least 1 dose of durvalumab on this study or enrolled on this study within 90 days of the last dose of durvalumab or durvalumab combination on the respective parent clinical study. All-cause mortality was reported for Full analysis set.
Arm/Group | Cohort 1: Durvalumab Continuation | Cohort 2: Durvalumab Restart | Cohort 3: No Restart of Durvalumab
All-Cause Mortality (participants affected / at risk) | 10/100 | 2/25 | 12/38
Serious Adverse Events (participants affected / at risk) | 23/100 | 0/7 | 0/2
Other Adverse Events (participants affected / at risk) | 72/100 | 1/7 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Durvalumab Continuation (N=100) | Cohort 2: Durvalumab Restart (N=7) | Cohort 3: No Restart of Durvalumab (N=2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Durvalumab Continuation (N=100) | Cohort 2: Durvalumab Restart (N=7) | Cohort 3: No Restart of Durvalumab (N=2)
Alanine aminotransferase increased (Investigations) | 7 (9) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 11 (17) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 8 (12) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 7 (14) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 8 (12) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 17 (17) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (10) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 8 (11) | 0 (0) | 0 (0)
Asthenia (General disorders) | 9 (9) | 0 (0) | 0 (0)
Fatigue (General disorders) | 11 (11) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 17 (19) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT04078152/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT04078152/SAP_001.pdf